CLINICAL TRIAL: NCT01243320
Title: In Vivo Assessment of Silver Biomaterial Nano-Toxicity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, mark munger, Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 40281
Record Dates: First submitted 2010-11-16; First posted 2010-11-18 (Estimated); Results first posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10ppm Oral Silver (Experimental): Oral Dose of 10ppm
  Interventions: Drug: 10ppm Oral Silver Particle
- 32ppm Oral Silver (Experimental): Oral Dose of 32ppm
  Interventions: Drug: 32ppm Oral Silver Particle

INTERVENTIONS:
Drug: 10ppm Oral Silver Particle — Silver nanoparticles at 10ppm
  Arms: 10ppm Oral Silver
Drug: 32ppm Oral Silver Particle — Silver nanoparticles at 32ppm
  Arms: 32ppm Oral Silver

SUMMARY:
Nanotechnology is the controlled generation and manipulation of matter in dimensions less than 100 nm. Silver has been used for its bactericidal properties. The investigators propose to study the American Biotech Laboratory 32 ppm silver solution over a 14-day period in human volunteers to determine the toxicity and to quantify cytochrome P450 enzyme effects of this solution.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be > 18-80 years old will be included.

Exclusion Criteria:

* Females of child-bearing potential, defined as women physically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means will be excluded unless they are using 2 barrier birth control methods (i.e., diaphragm, condom, intrauterine device, sponge or spermicide) or hormonal contraceptive method.
* Any female subject who is nursing will be excluded. Subject with has a history of heavy metal allergy (including silver) or a history of asthma or COPD or renal impairment defined by a creatinine clearance below 30 ml/min.
* Subjects with symptoms of an active upper respiratory infection at time of consent will also be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Munger, Pharm.D>, Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospital and Clinics, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Munger MA, Radwanski P, Hadlock GC, Stoddard G, Shaaban A, Falconer J, Grainger DW, Deering-Rice CE. In vivo human time-exposure study of orally dosed commercial silver nanoparticles. Nanomedicine. 2014 Jan;10(1):1-9. doi: 10.1016/j.nano.2013.06.010. Epub 2013 Jun 28. PMID 23811290

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Study had two dosing phases. All study participants were assigned the 10ppm Oral Silver and proceed to the 32 pm Oral Silver.
Period: 10ppm Oral Silver (3 Days)
Arm/Group | All Study Participants
Started | 36
Completed | 36
Not Completed | 0
Period: 10ppm Oral Silver (7 Days)
Arm/Group | All Study Participants
Started | 36
Completed | 36
Not Completed | 0
Period: 10ppm Oral Silver (14 Days)
Arm/Group | All Study Participants
Started | 36
Completed | 36
Not Completed | 0
Period: Washout (3 Days)
Arm/Group | All Study Participants
Started | 36
Completed | 36
Not Completed | 0
Period: 32ppm Oral Silver (14 Days)
Arm/Group | All Study Participants
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: 10 ppm Silver, then 32 ppm Silver
Arm/Group | All Study Participants
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 19

OUTCOME MEASURES:

1. Secondary Outcome: Change Systolic Blood Pressure
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: mmhg
Groups:
- 10ppm Oral Silver: ASAP Solution 10 ppm: Silver nanoparticles at 10ppm
- 32ppm Oral Silver: ASAP Solution 32 ppm Diluent: Silver nanoparticles at 32ppm
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
mmhg | 1.3 [-1.7 to 4.3] | -1.3 [-3.0 to 5.6]

2. Secondary Outcome: Mean Change in Diastolic Blood Pressure
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: mmhg
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
mmhg | -2.4 [-5.5 to 0.7] | -0.7 [-2.5 to 3.8]

3. Secondary Outcome: Mean Change in Heart Rate
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: bpm
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
bpm | -1.9 [-5.0 to 1.3] | -3.1 [-6.4 to 0.3]

4. Primary Outcome: Change in Sodium Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
mmol/L | -0.1 [-0.7 to 0.6] | 0.2 [-0.7 to 1.0]

5. Primary Outcome: Change in Potassium Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
mmol/L | -0.1 [-0.3 to 0.02] | -0.03 [-0.2 to 0.1]

6. Primary Outcome: Change in Chloride Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
mmol/L | -0.4 [-1.2 to 0.3] | 0.04 [-1.1 to 1.2]

7. Primary Outcome: Change in Carbon Dioxide Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
mmol/L | 0.5 [-0.5 to 1.6] | -0.04 [-1.1 to 1.0]

8. Primary Outcome: Change in Urea Nitrogen Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
mg/dL | -0.9 [-1.7 to -0.1] | 0.5 [-0.08 to 1.8]

9. Primary Outcome: Change In CreatinineBlood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
mg/dL | 0.01 [-0.02 to 0.03] | -0.02 [-0.04 to 0.01]

10. Primary Outcome: Change In Glucose Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
mg/dL | 3.6 [-1.6 to 8.7] | -0.7 [-4.2 to 2.9]

11. Primary Outcome: Change In Alkaline Phosphatase Blood Level
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: u/L
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
u/L | -1.4 [-3.9 to 1.1] | 2.0 [-1.0 to 5.0]

12. Primary Outcome: Change In Aspartate Aminotransferase Blood Level
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: u/L
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
u/L | -0.44 [-2.1 to 1.2] | 2.0 [-2.6 to 6.5]

13. Primary Outcome: Change In Alanine Aminotransferase Blood Level
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: u/L
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
u/L | -2.6 [-4.8 to -0.3] | 2.3 [-1.6 to 6.3]

14. Primary Outcome: Change In Total Protein Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
g/dL | -0.02 [-0.3 to 0.2] | 0.2 [-0.001 to 0.4]

15. Primary Outcome: Change In Total Bilirubin Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
mg/dL | -0.02 [-0.08 to 0.3] | -0.03 [-0.11 to 0.05]

16. Primary Outcome: Change in Albumin Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
g/dL | -0.07 [-0.1 to 0.0004] | 0.11 [-0.01 to 0.23]

17. Primary Outcome: Change In Calcium Blood Level
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
mg/dL | -0.1 [-0.2 to 0.04] | 0.1 [-0.003 to 0.2]

18. Primary Outcome: Change In White Blood Count Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: k/uL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
k/uL | -0.17 [-0.53 to 0.19] | -0.09 [-0.68 to 0.49]

19. Primary Outcome: Change In Red Blood Count Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: m/uL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
m/uL | -0.08 [-0.17 to -0.0001] | 0.06 [-0.03 to 0.14]

20. Primary Outcome: Change In Hemoglobin Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: gm/dL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
gm/dL | -0.2 [-0.4 to 0.03] | 0.1 [-0.2 to 0.4]

21. Primary Outcome: Change In Hematocrit Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
percent | -0.7 [-1.5 to 0.07] | 0.8 [-0.1 to 1.7]

22. Primary Outcome: Change In Mean Corpuscular Volume Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 days
Measure: Mean (95% Confidence Interval); unit: fL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
fL | 0.1 [-0.6 to 0.8] | 0.5 [-0.1 to 1.2]

23. Primary Outcome: Change In Mean Corpuscular Hemoglobin Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: pg
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
pg | 0.1 [-0.1 to 0.3] | -0.01 [-0.4 to 0.2]

24. Primary Outcome: Change In Mean Corpuscular Hemoglobin Concentration Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 days
Measure: Mean (95% Confidence Interval); unit: gm/dL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
gm/dL | 0.1 [-0.3 to 0.4] | -0.3 [-0.7 to 0.1]

25. Primary Outcome: Change In Platelet Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: k/uL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
k/uL | 5 [-6 to 15] | -4 [-16 to 8]

26. Primary Outcome: Change In Granulocytes Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
percent | -0.9 [-3.0 to 1.1] | -0.7 [-4.0 to 2.7]

27. Primary Outcome: Change In Lymphocytes Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
percent | 0.7 [-1.2 to 2.6] | 1.3 [-1.5 to 4.1]

28. Primary Outcome: Change In Monocytes Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
percent | -0.1 [-0.6 to 0.4] | -0.3 [-0.8 to 0.3]

29. Primary Outcome: Change in Basophils Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
percent | 0.04 [-0.1 to 0.2] | 0.001 [-0.1 to 0.1]

30. Primary Outcome: Change in Eosinophil Blood Levels
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
percent | -0.06 [-0.3 to 0.2] | -0.2 [-0.7 to 0.2]

31. Primary Outcome: Sputum Reactive Oxygen Species Change
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: uM
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
uM | 0.89 [-0.6 to 2.38] | -0.44 [-1.23 to 0.35]

32. Primary Outcome: Change to Interleukin-8 Receptor
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
ng/mL | 2.19 [-1.53 to 5.9] | 6.39 [-5.83 to 18.60]

33. Primary Outcome: Change to Interleukin-1 Alpha Receptor
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
ng/mL | -0.0005 [-0.0007 to 0.0006] | 0.0197 [-0.0014 to 0.0408]

34. Primary Outcome: Change to Interleukin-1 Beta Receptor
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
ng/mL | 0.017 [-0.011 to 0.044] | 0.027 [-0.058 to 0.112]

35. Primary Outcome: Change in Monocyte Chemotactic Protein 1
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
ng/mL | -0.028 [-0.084 to 0.028] | -0.004 [-0.026 to 0.017]

36. Primary Outcome: Change in Quinone Oxidoreductase 1 Gene
Description: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | 10ppm Oral Silver | 32ppm Oral Silver
Number analyzed (Participants) | 36 | 24
ng/mL | -0.0043 [-0.0115 to 0.029] | -0.0279 [-0.4671 to 0.4114]

ADVERSE EVENTS:
Groups:
- 10ppm Oral Solution; 32ppm Oral Solution: All participants received the 10ppm Silver, then progressed to the 32 ppm Silver.
Arm/Group | 10ppm Oral Solution | 32ppm Oral Solution
Serious Adverse Events (participants affected / at risk) | 1/36 | 0/24
Other Adverse Events (participants affected / at risk) | 0/36 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10ppm Oral Solution (N=36) | 32ppm Oral Solution (N=24)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No